CLINICAL TRIAL: NCT02433210
Title: A Clinical Study Comparing the Basic Performance and Blood Compatibility Characteristics of Nipro ELISIO-H, Gambro Polyflux Revaclear and Fresenius Optiflux Dialyzers
Brief Title: A Clinical Study Comparing Basic Performance and Hemocompatibility of 3 Different Dialyzers in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Nipro Medical Corporation (Industry); Dialysis Clinic, Inc. (Industry)
Responsible Party: Principal Investigator, Madhukar Misra, Professor of Clinical medicine, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2002150
Record Dates: First submitted 2014-12-16; First posted 2015-05-04 (Estimated); Results first posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Kidneys, Artificial

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (3):
- Solute Clearance (Active Comparator): Solute clearance at 60 minutes for urea, creatinine, phosphate, beta 2 microglobulin, and myoglobin will be determined three times for ELISIO-15H, Revaclear and Optiflux 160NR dialyzers at the 60 minute time point.
  Interventions: Device: ELISIO-15H; Device: Revaclear; Device: Optiflux
- Hemocompatibility (Active Comparator): Hemocompatibility will be determined using the markers C3a, C5a, thrombin/anti-thrombin complex and complete blood count with platelets will be determined one time for each dialyzer at session 2 and at time points 0, 15, 30, 60, and 240 minutes for ELISIO-15H, Revaclear and Optiflux 160NR dialyzers ..
  Interventions: Device: ELISIO-15H; Device: Revaclear; Device: Optiflux
- Solute removal rate (Active Comparator): Solute (urea, creatinine, phosphate, beta 2 macroglobulin, and myoglobin) removal rate will be determined time points 0 and 240 minutes for ELISIO-15H, Revaclear and Optiflux 160NR dialyzers .
  Interventions: Device: ELISIO-15H; Device: Revaclear; Device: Optiflux

INTERVENTIONS:
Device: ELISIO-15H — Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Other Names: dialyzer
Device: Revaclear — Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Other Names: Dialyzer
Device: Optiflux — Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Other Names: Dialyzer

SUMMARY:
The aim of the study is to confirm the safety and clinical effectiveness of Nipro ELISIO-15H and to compare its performance characteristics and hemocompatibility with those of the commercially available dialyzers in U.S.A., Gambro Polyflux Revaclear and Fresenius F160NRe.

10 stable patients will be dialyzed 3 times/week with each dialyzer over 3 weeks. Blood samples for several parameters will be collected during hemodialysis to assess the performance and hemocompatibility of the dialyzers under study. Data thus collected will be analyzed for comparison by standard statistical analysis.

DETAILED DESCRIPTION:
Current patients receiving dialysis treatment for end stage renal disease and who meet the inclusion/exclusion criteria will be entered into the study. These patients will continue on their standard dialysis regimen as stated in the clinics Standard Operating Procedures. Each patient will be studied for three weeks with each week starting with a dialyzer of a different manufacture but of comparable characteristics. Solute clearances and removal will be determined at each of the three dialysis sessions during the week. During session 2 of each week additional specimens will be taken to analyze for hemocompatibility. At the end of the study all clearances and the hemocompatibility markers for each dialyzer will be compared to one another as well as to the manufactures stated characteristics. Blood for the clearance and removal calculations will be taken at time 0, 60 minutes and 240 minutes. Blood for the hemocompatibility determinations will be taken at time 0, 15, 30, 60 and 240 minutes. Flow rates, anticoagulant therapy, erythropoietin therapy, venous and arterial pressures will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients 18 years or older
* Stable on hemodialysis for more than 3 months
* Stable hemoglobin between 11-12 g/dl
* Stable arteriovenous (AV) fistula vascular access
* Stable anticoagulation and ESA regimen
* No active infection
* Able to sign informed consent and able to participate in the study
* Medically stable

Exclusion Criteria:

* Participation in another study which may interfere with the planned study
* Active infection
* Medical conditions which may interfere with the study (cardiac, liver disease, Hepatitis)
* Allergy to dialyzer membrane materials e.g. polysulfone
* Patients which cannot tolerate Heparin
* Female who are pregnant or planning to be pregnant
* Problem with or allergy to anticoagulation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06; Primary Completion 2017-11-30 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Misra, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Dialysis Clinic Incorporated, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were pre-screened to determine if met inclusion/exclusion criteria by the study coordinator. If they met the criteria the primary investigator met with them explained the project and if interested he then consented them. Once consented the patient started the study on the following Monday.
Pre-assignment Details: There were no significant events. We didn't lose any consented patients prior to starting the study. There was no special preparation prior to start of study other than inclusion/exclusion criteria which took place prior to consent.
Groups:
- Experimental: ELISIO, Then Revaclear, Then Optiflux: This group will start week one with the ELISIO dialyzer, followed by the Revaclear dialyzer in week two and in the third finish with the Optiflux dialyzer. Each patient will undergo three successive hemodialysis sessions during each week following their established regimen.
- Experimental: Revaclear, Then Optiflux, Then ELISIO: This group will start week one with the Revaclear dialyzer, followed by the Optiflux dialyzer in week two and finish with the ELISIO dialyzer in week three. . Each patient will undergo three successive hemodialysis sessions during each week following their established regimen.
- Experimental: Optiflux, Then ELISIO, Then Revaclear: This group will start with the Optiflux dialyzer in week one, followed by the ELISIO dialyzer in week two and finish with the Revaclear dialyzer in week three. Each patient will undergo three successive hemodialysis sessions during each week following their established regimen.
Period: Overall Study
Arm/Group | Experimental: ELISIO, Then Revaclear, Then Optiflux | Experimental: Revaclear, Then Optiflux, Then ELISIO | Experimental: Optiflux, Then ELISIO, Then Revaclear
Started | 5 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant was removed by the PI when it was determined that he had had a procedure to the fistula during the study period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: ELISIO, Then Revaclear, Then Optiflux | Experimental: Revaclear, Then Optiflux, Then ELISIO | Experimental: Optiflux, Then ELISIO, Then Revaclear | Total
Number analyzed (Participants) | 4 | 3 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 7
  >=65 years | 2 | 0 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was recorded at the time the patient started the study.
  years | 60.5 (14.8) | 53.6 (3.9) | 56.3 (7.8) | 57.2 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 3 | 3 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 2 | 1 | 1 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Clearance and Solute Removal Characteristics of Dialyzers
Description: Clearances of small, middle and large molecular weight solutes will be measured at 60 minute time point utilizing urea, creatinine, beta 2 microglobulin, phosphate and myoglobin. Dialyzer clearance is calculated as follows: 60 minute clearance:((([S]60'Art - [S]60'Ven) / [S]60'Art) * Qb) where [S] = solute concentration; Qb = blood flow rate. S
Time Frame: During each of the three weekly dialysis sessions measurements of urea were made at the 60 minute time point for each patient in the study. At the end of the study all measurements were summed for each of the three dialyzers.
Measure: Mean (Standard Deviation); unit: milliliters per minute (ml/min)
Groups:
- BUN Clearance Optiflux: Solute clearance at 60 minutes for urea
  ELISIO-15H: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Revaclear: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Optiflux: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
- BUN Clearance Revaclear; BUN Clearance Elisio: Solute clearance at 60 minutes for urea. ELISIO-15H: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Revaclear: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Optiflux: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
- Creatinine Clearance Optiflux: Solute clearance at 60 minutes for creatinine.
- Creatinine Clearance Revaclear: Solute clearance at 60 minutes for creatinine.
  ELISIO-15H: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Revaclear: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Optiflux: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
- Creatinine Clearance ELISIO: Solute clearance at 60 minutes for creatinine,
  ELISIO-15H: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Revaclear: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
  Optiflux: Each patient to undergo 3 successive hemodialysis/week with this dialyzer.
- Phosphate Clearance Optiflux; Phosphate Clearance Revaclear; Phosphate Clearance Elisio: Phosphate clearance at 60 minutes
- Beta 2 Microglobulin Revaclear; Beta 2 Microglobulin Optiflux; Beta 2 Microglobulin ELISIO: Beta 2 microglobulin clearance at 60 minutes
- Myoglobin Clearance Optiflux; Myoglobin Clearance Revaclear; Myoglobin Clearance ELISIO: Myoglobin clearance at 60 minutes.
Arm/Group | BUN Clearance Optiflux | BUN Clearance Revaclear | BUN Clearance Elisio | Creatinine Clearance Optiflux | Creatinine Clearance Revaclear | Creatinine Clearance ELISIO | Phosphate Clearance Optiflux | Phosphate Clearance Revaclear | Phosphate Clearance Elisio | Beta 2 Microglobulin Revaclear | Beta 2 Microglobulin Optiflux | Beta 2 Microglobulin ELISIO | Myoglobin Clearance Optiflux | Myoglobin Clearance Revaclear | Myoglobin Clearance ELISIO
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
milliliters per minute (ml/min)
  Session 1 | 354.1 (48) | 340.4 (72.5) | 361.8 (51) | 271.8 (65.2) | 295.9 (53.7) | 298.4 (49.3) | 309.8 (71) | 324.8 (60.5) | 333.1 (48.3) | 137.6 (38.7) | 57.2 (41.5) | 169.1 (59.6) | -7.1 (29) | 24.5 (57.6) | 33.4 (47.4)
  Session 2 | 336.2 (57.4) | 352.8 (40.1) | 356.3 (44.1) | 256.7 (78.6) | 297.6 (39.9) | 293.4 (37) | 306.4 (43) | 324.7 (45.3) | 277 (90.3) | 144 (26.8) | 63 (49.7) | 165.7 (51.5) | -2.6 (26.4) | 32.6 (53.5) | 19.1 (64.3)
  Session 3 | 331.9 (62.9) | 318.8 (69.4) | 355.7 (58.3) | 277.8 (59.2) | 275.5 (39.2) | 296.6 (33.3) | 296.6 (69.7) | 276.6 (100.9) | 330.4 (47.9) | 149.6 (28) | 61.4 (24.7) | 136.4 (90.3) | -8.6 (12.6) | 62.1 (108.2) | 45.5 (40)
Statistical Analysis 1: Comparison: Beta 2 Microglobulin Revaclear vs Beta 2 Microglobulin Optiflux; Session 1 clearance beta 2 microglobilin Optiflux vs Revaclear; Test type: Superiority; p < 0.001, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; Shapiro-Wilk test for Normality and equal variance was used. If data failed either non-parametric Mann-Whitney Rank sum test was used
Statistical Analysis 2: Comparison: Beta 2 Microglobulin Optiflux vs Beta 2 Microglobulin ELISIO; Session 1 Clearance beta 2 microglobulin Optiflux vs ELISIO; Test type: Superiority; p < 0.001, t-test, 2 sided — The p value is not adjusted for multiple comparisons and a p<0.05 is considered significant; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Beta 2 Microglobulin Revaclear vs Beta 2 Microglobulin ELISIO; Session 1 clearance beta 2 microglobulin Revaclear vs ELISIO; Test type: Superiority; p = 0.178, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Myoglobin Clearance Optiflux vs Myoglobin Clearance Revaclear; Session 1 Clearance of myoglobin Optiflux vs Revaclear; Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney) — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Myoglobin Clearance Optiflux vs Myoglobin Clearance ELISIO; Session 1 Clearance of myoglobin Optiflux vs ELISIO; Test type: Superiority; p = 0.033, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Beta 2 Microglobulin Optiflux vs Beta 2 Microglobulin ELISIO vs Myoglobin Clearance Revaclear vs Myoglobin Clearance ELISIO; Session 1 Clearance of myoglobin Revaclear vs ELISIO; Test type: Superiority; p = 0.935, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: BUN Clearance Optiflux vs BUN Clearance Revaclear; Session 2 Clearance of urea nitrogen Optiflux vs Revaclaer; Test type: Superiority; p = 0.463, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: BUN Clearance Optiflux vs BUN Clearance Elisio; Session 2 Clearance of urea nitrogen Optiflux vs ELISIO; Test type: Superiority; p = 0.392, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: BUN Clearance Revaclear vs BUN Clearance Elisio; Session 2 Clearance urea nitrogen Revaclear vs ELISIO; Test type: Superiority; p = 0.597, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Creatinine Clearance Optiflux vs Creatinine Clearance Revaclear; Session 2 Clearance of creatinine Optiflux vs Revaclear; Test type: Superiority; p = 0.162, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Creatinine Clearance Optiflux vs Creatinine Clearance ELISIO; Session 2 Clearance of creatinine Optiflux vs ELISIO; Test type: Superiority; p = 0.186, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: BUN Clearance Optiflux vs BUN Clearance Revaclear; Session 1 Urea nitrogen clearance Optiflux vs Revaclear; Test type: Superiority — No Significant difference; p = 0.624, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: BUN Clearance Optiflux vs BUN Clearance Elisio; Session 1 Urea nitrogen clearance Optiflux vs ELISIO; Test type: Superiority; p = 0.732, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: BUN Clearance Revaclear vs BUN Clearance Elisio; Session 1 Urea Nitrogen clearance Revaclear vs Optiflux; Test type: Superiority; p = 0.427, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: BUN Clearance Revaclear vs Creatinine Clearance Optiflux; Session 1 Creatinine clearance Optiflux vs Revaclear; Test type: Superiority; p = 0.379, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Creatinine Clearance Optiflux vs Creatinine Clearance ELISIO; Session 1 Creatinine clearance Optiflux vs ELISIO; Test type: Superiority; p = 0.318, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Creatinine Clearance Revaclear vs Creatinine Clearance ELISIO; Session 1 Creatinine clearance Revaclear vs ELISIO; Test type: Superiority; p = 0.914, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Phosphate Clearance Optiflux vs Phosphate Clearance Revaclear; Session 1 Phosphate clearance Optiflux vs Revaclear; Test type: Superiority; p = 0.623, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Phosphate Clearance Optiflux vs Phosphate Clearance Elisio; Session 1 Phosphate clearance Optiflux vs ELISIO; Test type: Superiority; p = 0.403, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Phosphate Clearance Revaclear vs Phosphate Clearance Elisio; Session 1 Phosphate clearance Revaclear vs ELISIO; Test type: Superiority; p = 0.850, Wilcoxon (Mann-Whitney); Shapiro-Wilk test for Normality and an equal variance was used. If data failed either, non-parametric Mann-Whitney Rank sum test was used
Statistical Analysis 21: Comparison: Creatinine Clearance Revaclear vs Creatinine Clearance ELISIO; Session 2 Clearance of creatinine Revaclear vs ELISIO; Test type: Superiority; p = 0.815, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 22: Comparison: Phosphate Clearance Optiflux vs Phosphate Clearance Revaclear; Session 2 Clearance of Phosphate Optiflux vs Revaclear; Test type: Superiority; p = 0.367, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 23: Comparison: Phosphate Clearance Optiflux vs Phosphate Clearance Elisio; Session 2 Clearance of phosphate Optiflux vs Elisio; Test type: Superiority; p = 0.821, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 20]
Statistical Analysis 24: Comparison: Phosphate Clearance Revaclear vs Phosphate Clearance Elisio; Session 2 Clearance phosphate Revaclear vs ELISIO; Test type: Superiority; p = 0.364, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 20]
Statistical Analysis 25: Comparison: Beta 2 Microglobulin Revaclear vs Beta 2 Microglobulin Optiflux; Session 2 Clearance of beta 2 microglobulin Optiflux vs Revaclear; Test type: Superiority; p < 0.001, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 26: Comparison: Beta 2 Microglobulin Optiflux vs Beta 2 Microglobulin ELISIO; Session 2 Clearance of beta 2 microglobulin Optiflux vs ELISIO; Test type: Superiority; p < 0.001, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 27: Comparison: Beta 2 Microglobulin Revaclear vs Beta 2 Microglobulin ELISIO; Session 2 Clearance of beta 2 microglobulin Revaclear vs ELISIO; Test type: Superiority; p = 0.254, t-test, 2 sided
Statistical Analysis 28: Comparison: Myoglobin Clearance Optiflux vs Myoglobin Clearance Revaclear; Session 2 Clearance of myoglobin Optiflux vs Revaclear; Test type: Superiority; p = 0.079, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 29: Comparison: Myoglobin Clearance Optiflux vs Myoglobin Clearance ELISIO; Session 2 Clearance of myoglobin Optiflux vs ELISIO; Test type: Superiority; p = 0.086, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 20]
Statistical Analysis 30: Comparison: Myoglobin Clearance Revaclear vs Myoglobin Clearance ELISIO; Session 2 Clearance myoglobin Revaclear vs ELISIO; Test type: Superiority; p = 0.888, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 31: Comparison: BUN Clearance Optiflux vs BUN Clearance Revaclear; Session 3 Clearance of urea nitrogen Optiflux vs Revaclear; Test type: Superiority; p = 0.663, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 32: Comparison: BUN Clearance Optiflux vs BUN Clearance Elisio; Session 3 Clearance of urea nitrogen Optiflux vs ELISIO; Test type: Superiority; p = 0.391, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 33: Comparison: BUN Clearance Revaclear vs BUN Clearance Elisio; Session 3 Clearance of urea nitrogen Revaclear vs ELISIO; Test type: Superiority; p = 0.214, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 34: Comparison: Creatinine Clearance Optiflux vs Creatinine Clearance Revaclear; Session 3 Clearance of creatinine Optiflux vs Revaclear; Test type: Superiority; p = 0.918, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 35: Comparison: Creatinine Clearance Optiflux vs Creatinine Clearance ELISIO; Session 3 Clearance of creatinine Optiflux vs ELISIO; Test type: Superiority; p = 0.394, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 36: Comparison: Creatinine Clearance Revaclear vs Creatinine Clearance ELISIO; Session 3 Clearance of creatinine Revaclear vs ELISIO; Test type: Superiority; p = 0.211, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 37: Comparison: Phosphate Clearance Optiflux vs Phosphate Clearance Elisio; Session 3 Clearance of phosphate Optiflux vs ELISIO; Test type: Superiority; p = 0.222, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 38: Comparison: Phosphate Clearance Revaclear vs Phosphate Clearance Elisio; Session 3 Clearances of phosphate Revaclear vs ELISIO; Test type: Superiority; p = 0.162, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 20]
Statistical Analysis 39: Comparison: Beta 2 Microglobulin Revaclear vs Beta 2 Microglobulin Optiflux; Session 3 Clearance of beta 2 microglobulin Optiflux vs Revaclear; Test type: Superiority; p < 0.001, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 40: Comparison: Beta 2 Microglobulin Optiflux vs Beta 2 Microglobulin ELISIO; Session 3 Clearances of beta 2 microglobulin Optiflux vs ELISIO; Test type: Superiority; p = 0.025, Wilcoxon (Mann-Whitney) — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 41: Comparison: Beta 2 Microglobulin Revaclear vs Beta 2 Microglobulin ELISIO; Session 3 Clearance of beta 2 microglobulin Revaclear vs ELISIO; Test type: Superiority; p = 0.903, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 20]
Statistical Analysis 42: Comparison: Myoglobin Clearance Optiflux vs Myoglobin Clearance Revaclear; Session 3 Clearances of myoglobin Optiflux vs Revaclear; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney) — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 43: Comparison: Myoglobin Clearance Optiflux vs Myoglobin Clearance ELISIO; Session 3 Clearance of myoglobin Optiflux vs ELISIO; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 44: Comparison: Myoglobin Clearance Revaclear vs Myoglobin Clearance ELISIO; Session 3 Clearance of myoglobin Revaclear vs ELISIO; Test type: Superiority; p = 0.472, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 20]

2. Primary Outcome: Hemocompatibility as Shown by C5a for Optiflux, Revaclear, and ELISIO Hemodialysis Dialyzers of Dialyzers
Description: The molecules monitored will be C5a, thrombin/anti-thrombin complex and a complete blood count with platelets.
Time Frame: Once a week during the second of the three weekly sessions specimens will be taken at time points 0, 15, 30, 60 and 240 minutes. Measurements, all patients, were summed for each dialyzer type by time period.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Groups:
- % Change in C5a at 15 Minutes Optiflux: Percent change from Baseline at 15 minutes C5a, .
- % Change in C5a at 15 Minutes Revaclear; %Change in C5a at 15 Minutes ELISIO: Percent change from baseline at 15 minutes for C5a.
- % Change in C5a at 30 Minutes Optiflux; % Change in C5a at 30 Minutes Revaclear; % Change in C5a at 30 Minutes ELISIO: Percent change from baseline at 30 minutes for C5a.
- % Change in C5a at 60 Minutes Optiflux; % Change in C5a at 60 Minutes Revaclear; % Change in C5a at 60 Minutes ELISIO: Percent change from baseline at 60 minutes for C5a.
- % Change in C5a at 240 Minutes Optiflux; % Change in C5a at 240 Minutes Revaclear; % Change in C5a at 240 Minutes ELISIO: Percent change from baseline at 240 minutes for C5a.
Arm/Group | % Change in C5a at 15 Minutes Optiflux | % Change in C5a at 15 Minutes Revaclear | %Change in C5a at 15 Minutes ELISIO | % Change in C5a at 30 Minutes Optiflux | % Change in C5a at 30 Minutes Revaclear | % Change in C5a at 30 Minutes ELISIO | % Change in C5a at 60 Minutes Optiflux | % Change in C5a at 60 Minutes Revaclear | % Change in C5a at 60 Minutes ELISIO | % Change in C5a at 240 Minutes Optiflux | % Change in C5a at 240 Minutes Revaclear | % Change in C5a at 240 Minutes ELISIO
Number analyzed (Participants) | 10 | 8 | 10 | 10 | 8 | 10 | 9 | 8 | 10 | 10 | 8 | 10
Percent change from baseline | 8.5 (28.0) | -5.1 (26.8) | -4.5 (15.4) | 11.2 (17.8) | 7.5 (25.3) | -1.1 (19.6) | -17.7 (22.8) | -9.8 (22.7) | -6.1 (35.4) | 15.9 (15.6) | -6.6 (14.3) | 1 (31.7)
Statistical Analysis 1: Comparison: % Change in C5a at 15 Minutes Optiflux vs % Change in C5a at 15 Minutes Revaclear; Test type: Superiority; p = 0.216, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 2: Comparison: % Change in C5a at 15 Minutes Optiflux vs %Change in C5a at 15 Minutes ELISIO; Test type: Superiority — No significant difference; p = 0.216, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 3: Comparison: % Change in C5a at 15 Minutes Revaclear vs %Change in C5a at 15 Minutes ELISIO; Test type: Superiority — No significant difference; p = 0.952, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 4: Comparison: % Change in C5a at 30 Minutes Optiflux vs % Change in C5a at 30 Minutes Revaclear; Test type: Superiority — No Significant difference; p = 0.714, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 5: Comparison: % Change in C5a at 30 Minutes Optiflux vs % Change in C5a at 30 Minutes ELISIO; Test type: Superiority; p = 0.156, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 6: Comparison: % Change in C5a at 30 Minutes Revaclear vs % Change in C5a at 30 Minutes ELISIO; Test type: Superiority; p = 0.427, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 7: Comparison: % Change in C5a at 60 Minutes Optiflux vs % Change in C5a at 60 Minutes Revaclear; No significant difference; Test type: Superiority; p = 0.487, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 8: Comparison: % Change in C5a at 60 Minutes Optiflux vs % Change in C5a at 60 Minutes ELISIO; No significant difference; Test type: Superiority — Failed normality test; p = 0.111, Wilcoxon (Mann-Whitney) — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; The difference in the median values between the two groups is not > enough to exclude that the difference is due to random sampling variability
Statistical Analysis 9: Comparison: % Change in C5a at 60 Minutes Revaclear vs % Change in C5a at 60 Minutes ELISIO; No significant difference; Test type: Superiority — Failed normality test; p = 0.198, Wilcoxon (Mann-Whitney) — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 10: Comparison: % Change in C5a at 240 Minutes Optiflux vs % Change in C5a at 240 Minutes Revaclear; Showed a significant difference; Test type: Superiority; p = 0.007, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 11: Comparison: % Change in C5a at 240 Minutes Optiflux vs % Change in C5a at 240 Minutes ELISIO; No significant difference; Test type: Superiority; p = 0.202, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 12: Comparison: % Change in C5a at 240 Minutes Revaclear vs % Change in C5a at 240 Minutes ELISIO; No significant difference; Test type: Superiority; p = 0.540, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]

3. Primary Outcome: Hemocompatibility as Shown by Thrombin/Antithrombin Complex for Optiflux, Revaclear, and ELISIO Hemodialysis Dialyzers.
Description: Measure of the % change from Baseline for the hemocompatibility marker Thrombin/Antithrombin complex for the Optiflux, Revaclear, and ELISIO dialyzers.
Time Frame: Once a week during the second of the three weekly sessions specimens will be taken at the 60 and 240 minutes timepoints. Measurements for all patients were summed for each dialyzer type by time period for analysis..
Measure: Mean (Standard Deviation); unit: % Change from Baseline
Groups:
- Thrombin/Anti-Thrombin 60 Minutes Optiflux: This is the percent change from baseline at 60 minutes for Thrombin/Anti-Thrombin Complex in the Optiflux dialyzer.
- Thrombin/Antithrombin 60 Minutes Revaclear: This is the percent change from Baseline at 60 minutes for Thrombin/Antithrombin Complex in the Revaclear Dialyzer.
- Thrombin/Antithrombin 60 Minutes ELISIO: This is the percent change from baseline at 60 minutes for Thrombin/Antithrombin Complex in ELISIO dialyzers.
- Thrombin/Antithrombin 240 Minutes Optiflux: This is the percent change from baseline at 240 minutes for Thrombin/Antithrombin Complex in Optiflux dialyzers.
- Thrombin/Antithrombin 240 Minutes Revaclear: This is the percent of change from baseline at 240 minutes for Thrombin/Antithrombin Complex in Revaclear dialyzers.
- Thrombin/Antithrombin 240 Minutes ELISIO: This is the percent change from baseline at 240 minutes for Thrombin/Antithrombin Complex in ELISIO dialyzers.
Arm/Group | Thrombin/Anti-Thrombin 60 Minutes Optiflux | Thrombin/Antithrombin 60 Minutes Revaclear | Thrombin/Antithrombin 60 Minutes ELISIO | Thrombin/Antithrombin 240 Minutes Optiflux | Thrombin/Antithrombin 240 Minutes Revaclear | Thrombin/Antithrombin 240 Minutes ELISIO
Number analyzed (Participants) | 7 | 9 | 6 | 8 | 9 | 9
% Change from Baseline | 35.8 (99.5) | -16.4 (44.3) | 52.7 (50.4) | 895.3 (755.0) | 474.7 (393.9) | 545.2 (573.1)
Statistical Analysis 1: Comparison: Thrombin/Anti-Thrombin 60 Minutes Optiflux vs Thrombin/Antithrombin 60 Minutes Revaclear; Test type: Superiority; p = 0.204, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Thrombin/Anti-Thrombin 60 Minutes Optiflux vs Thrombin/Antithrombin 60 Minutes ELISIO; Test type: Superiority; p = 0.234, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Thrombin/Antithrombin 60 Minutes Revaclear vs Thrombin/Antithrombin 60 Minutes ELISIO; Test type: Superiority; p = 0.015, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the <0.050 level; Shapiro-Wilk test for Normality and an equal variance was used. If data failed either then the non-parametric Mann-Whitney Rank Sum Test was used
Statistical Analysis 4: Comparison: Thrombin/Antithrombin 240 Minutes Optiflux vs Thrombin/Antithrombin 240 Minutes Revaclear; Test type: Superiority; p = 0.413, Wilcoxon (Mann-Whitney) — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 5: Comparison: Thrombin/Antithrombin 240 Minutes Optiflux vs Thrombin/Antithrombin 240 Minutes ELISIO; Test type: Superiority; p = 0.314, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 6: Comparison: Thrombin/Antithrombin 240 Minutes Revaclear vs Thrombin/Antithrombin 240 Minutes ELISIO; Test type: Superiority; p = 0.769, t-test, 2 sided — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]

4. Primary Outcome: Hemocompatibility as Shown by Hematocrit for Optiflux, Revaclear, and ELISIO Hemodialysis Dialyzers
Description: Measure of the % change from Baseline for the hemocompatibility marker Hematocrit for the Optiflux, Revaclear, and ELISIO dialyzers.
Time Frame: Once a week during the second of three weekly sessions samples will be taken at the 0, 15, 30, 60, and 240 minute timepoints. Measurements for all patients were summed for each dialyzer type by time period for analysis.
Measure: Mean (Standard Deviation); unit: Percent change from baseline.
Groups:
- Hematocrit 15 Minutes Optiflux: % Change in Hematocrit at 15 minutes for Optiflux.
- Hematocrit 15 Minutes Revaclear: % Change in Hematocrit at 15 minutes for Revaclear.
- Hematocrit 15 Minutes ELISIO: % Change in Hematocrit at 15 minutes for ELISIO.
- Hematocrit 30 Minutes Optiflux: % Change in Hematocrit at 30 minutes for Optiflux.
- Hematocrit 30 Minutes Revaclear: % Change in Hematocrit at 30 minutes for Revaclear.
- Hematocrit 30 Minutes ELISIO: % Change in Hematocrit at 30 minutes for ELISIO.
- Hematocrit 60 Minutes Optiflux: % Change in Hematocrit at 60 minutes for Optiflux.
- Hematocrit 60 Minutes Revaclear: % Change in Hematocrit at 60 minutes for Revaclear.
- Hematocrit 60 Minutes ELISIO: % Change in Hematocrit at 60 minutes for ELISIO.
- Hematocrit 240 Minutes Optiflux: % Change in Hematocrit at 240 minutes for Optiflux.
- Hematocrit 240 Minutes Revaclear: % Change in Hematocrit at 240 minutes for Revaclear.
- Hematocrit 240 Minutes ELISIO: % Change in Hematocrit at 240 minutes for ELISIO.
Arm/Group | Hematocrit 15 Minutes Optiflux | Hematocrit 15 Minutes Revaclear | Hematocrit 15 Minutes ELISIO | Hematocrit 30 Minutes Optiflux | Hematocrit 30 Minutes Revaclear | Hematocrit 30 Minutes ELISIO | Hematocrit 60 Minutes Optiflux | Hematocrit 60 Minutes Revaclear | Hematocrit 60 Minutes ELISIO | Hematocrit 240 Minutes Optiflux | Hematocrit 240 Minutes Revaclear | Hematocrit 240 Minutes ELISIO
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 10 | 9 | 9 | 10 | 9 | 9 | 10 | 9
Percent change from baseline. | -5.8 (6.2) | -3.2 (6.1) | -4.2 (4.4) | -3.8 (3.7) | -2.1 (5.3) | -1.0 (5.6) | -1.8 (4.0) | -3.0 (6.7) | 0.03 (5.6) | 0.8 (7.0) | 1.9 (6.5) | 2.0 (8.3)
Statistical Analysis 1: Comparison: Hematocrit 15 Minutes Optiflux vs Hematocrit 15 Minutes Revaclear; Test type: Superiority; p = 0.376, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 2: Comparison: Hematocrit 15 Minutes Optiflux vs Hematocrit 15 Minutes ELISIO; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney) — The p value was not adjusted for multiple comparisons and the difference was considered significant at the p<0.05 level; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 3: Comparison: Hematocrit 15 Minutes Revaclear vs Hematocrit 15 Minutes ELISIO; Test type: Superiority; p = 0.713, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 20]
Statistical Analysis 4: Comparison: Hematocrit 30 Minutes Optiflux vs Hematocrit 30 Minutes Revaclear; Test type: Superiority; p = 0.424, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 5: Comparison: Hematocrit 30 Minutes Optiflux vs Hematocrit 30 Minutes ELISIO; Test type: Superiority; p = 0.230, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 6: Comparison: Hematocrit 30 Minutes Revaclear vs Hematocrit 30 Minutes ELISIO; Test type: Superiority; p = 0.678, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 7: Comparison: Hematocrit 60 Minutes Optiflux vs Hematocrit 60 Minutes ELISIO; Test type: Superiority; p = 0.643, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 8: Comparison: Hematocrit 60 Minutes Optiflux vs Hematocrit 60 Minutes ELISIO; Test type: Superiority; p = 0.430, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 9: Comparison: Hematocrit 60 Minutes Revaclear vs Hematocrit 60 Minutes ELISIO; Test type: Superiority; p = 0.295, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 10: Comparison: Hematocrit 240 Minutes Optiflux vs Hematocrit 240 Minutes Revaclear; Test type: Superiority; p = 0.723, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 11: Comparison: Hematocrit 240 Minutes Optiflux vs Hematocrit 240 Minutes ELISIO; Test type: Superiority; p = 0.749, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 12: Comparison: Hematocrit 240 Minutes Revaclear vs Hematocrit 240 Minutes ELISIO; Test type: Superiority; p = 0.967, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 20]

5. Primary Outcome: Hemocompatibility as Shown by Hemoglobin for Optiflux, Revaclear, and ELISIO Hemodialysis Dialyzers
Description: Measure of the % change from Baseline for the hemocompatibility marker Hemoglobin for the Optiflux, Revaclear, and ELISIO dialyzers.
Time Frame: Once a week during the second of the three weekly sessions samples will be taken at the 0, 15, 30, 60 and 240 minutes time points. Measurements for all patients were summed for each dialyzer type and time point for analysis.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Groups:
- % Change in Hemoglobin at 15 Minutes Optiflux; % Change in Hemoblobin at 15 Minutes Revaclear; % Change in Hemoblobin at 15 Minutes ELISIO: Percent change from baseline at 15 minutes for hemoglobin.
- % Change in Hemoblobin at 30 Minutes Optiflux; % Change in Hemoblobin at 30 Minutes Revaclear; % Change in Hemoblobin at 30 Minutes ELISIO: Percent change from baseline at 30 minutes for hemoglobin.
- % Change in Hemoblobin at 60 Minutes Optiflux; % Change in Hemoblobin at 60 Minutes Revaclear; % Change in Hemoblobin at 60 Minutes ELISIO: Percent change from baseline at 60 minutes for hemoglobin.
- % Change in Hemoblobin at 240 Minutes Optiflux; % Change in Hemoblobin at 240 Minutes Revaclear; % Change in Hemoblobin at 240 Minutes ELISIO: Percent change from baseline at 240 minutes for hemoglobin.
Arm/Group | % Change in Hemoglobin at 15 Minutes Optiflux | % Change in Hemoblobin at 15 Minutes Revaclear | % Change in Hemoblobin at 15 Minutes ELISIO | % Change in Hemoblobin at 30 Minutes Optiflux | % Change in Hemoblobin at 30 Minutes Revaclear | % Change in Hemoblobin at 30 Minutes ELISIO | % Change in Hemoblobin at 60 Minutes Optiflux | % Change in Hemoblobin at 60 Minutes Revaclear | % Change in Hemoblobin at 60 Minutes ELISIO | % Change in Hemoblobin at 240 Minutes Optiflux | % Change in Hemoblobin at 240 Minutes Revaclear | % Change in Hemoblobin at 240 Minutes ELISIO
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 10 | 9 | 9 | 10 | 9 | 9 | 10 | 9
Percent Change from Baseline | -2.3 (2.0) | -1.8 (3.0) | -2.3 (1.6) | -2.2 (1.9) | -1.1 (2.7) | -2.7 (2.1) | -0.9 (2.7) | -1.2 (2.8) | -1.7 (2.3) | 2.3 (5.2) | 4.3 (4.3) | 2.4 (4.6)
Statistical Analysis 1: Comparison: % Change in Hemoglobin at 15 Minutes Optiflux vs % Change in Hemoblobin at 15 Minutes Revaclear; Test type: Superiority; p = 0.670, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 2: Comparison: % Change in Hemoglobin at 15 Minutes Optiflux vs % Change in Hemoblobin at 15 Minutes ELISIO; Test type: Superiority; p = 0.993, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 3: Comparison: % Change in Hemoblobin at 15 Minutes Revaclear vs % Change in Hemoblobin at 15 Minutes ELISIO; Test type: Superiority; p = 0.650, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 4: Comparison: % Change in Hemoblobin at 30 Minutes Optiflux vs % Change in Hemoblobin at 30 Minutes Revaclear; Test type: Superiority; p = 0.299, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 5: Comparison: % Change in Hemoblobin at 30 Minutes Optiflux vs % Change in Hemoblobin at 30 Minutes ELISIO; Test type: Superiority; p = 0.659, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 6: Comparison: % Change in Hemoblobin at 30 Minutes Revaclear vs % Change in Hemoblobin at 30 Minutes ELISIO; Test type: Superiority; p = 0.176, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 7: Comparison: % Change in Hemoblobin at 60 Minutes Optiflux vs % Change in Hemoblobin at 60 Minutes Revaclear; Test type: Superiority; p = 0.853, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 8: Comparison: % Change in Hemoblobin at 60 Minutes Optiflux vs % Change in Hemoblobin at 60 Minutes ELISIO; Test type: Superiority; p = 0.494, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 9: Comparison: % Change in Hemoblobin at 60 Minutes Revaclear vs % Change in Hemoblobin at 60 Minutes ELISIO; Test type: Superiority; p = 0.631, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 10: Comparison: % Change in Hemoblobin at 240 Minutes Optiflux vs % Change in Hemoblobin at 240 Minutes Revaclear; Test type: Superiority; p = 0.370, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 11: Comparison: % Change in Hemoblobin at 240 Minutes Optiflux vs % Change in Hemoblobin at 240 Minutes ELISIO; Test type: Superiority; p = 0.950, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 12: Comparison: % Change in Hemoblobin at 240 Minutes Revaclear vs % Change in Hemoblobin at 240 Minutes ELISIO; Test type: Superiority; p = 0.377, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]

6. Primary Outcome: Hemocompatibility as Shown by White Cell Count for Optiflux, Revaclear, and ELISIO Hemodialysis Dialyzers
Description: Measure of the % change from Baseline for the hemocompatibility marker White Cell Count for the Optiflux, Revaclear, and ELISIO dialyzers.
Time Frame: Once a week during the second of the three weekly sessions samples will be taken at the 0, 15, 30, 60 and 240 minutes time periods. All measurements for all patients were summed for each dialyzer type and time point.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Groups:
- % Change in White Cell Count at 15 Minutes Optiflux: Percent change from baseline at 15 minutes for hemoglobin.
- % Change in White Cell Count at 15 Minutes Revaclear; % Change in White Cell Count at 15 Minutes ELISIO: Percent change from baseline at 15 minutes for white cell count.
- % Change in White Cell Count at 30 Minutes Optiflux; % Change in White Cell Count at 30 Minutes Revaclear; % Change in White Cell Count at 30 Minutes ELISIO: Percent change from baseline at 30 minutes for white cell count.
- % Change in White Cell Count at 60 Minutes Optiflux; % Change in White Cell Count at 60 Minutes Revaclear; % Change in White Cell Count at 60 Minutes ELISIO: Percent change from baseline at 60 minutes for white cell count.
- % Change in White Cell Count at 240 Minutes Optiflux; % Change in White Cell Count at 240 Minutes Revaclear; % Change in White Cell Count at 240 Minutes ELISIO: Percent change from baseline at 240 minutes for white cell count.
Arm/Group | % Change in White Cell Count at 15 Minutes Optiflux | % Change in White Cell Count at 15 Minutes Revaclear | % Change in White Cell Count at 15 Minutes ELISIO | % Change in White Cell Count at 30 Minutes Optiflux | % Change in White Cell Count at 30 Minutes Revaclear | % Change in White Cell Count at 30 Minutes ELISIO | % Change in White Cell Count at 60 Minutes Optiflux | % Change in White Cell Count at 60 Minutes Revaclear | % Change in White Cell Count at 60 Minutes ELISIO | % Change in White Cell Count at 240 Minutes Optiflux | % Change in White Cell Count at 240 Minutes Revaclear | % Change in White Cell Count at 240 Minutes ELISIO
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 10 | 9 | 9 | 10 | 9 | 9 | 10 | 9
Percent Change from Baseline | -8.1 (8.0) | -5.8 (7.4) | -10.1 (7.5) | -5.5 (6.5) | -0.8 (6.2) | -2.9 (8.2) | -3.9 (6.2) | -2.4 (5.1) | -3.8 (5.3) | -3.2 (12.4) | 2.9 (9.5) | -0.06 (6.4)
Statistical Analysis 1: Comparison: % Change in White Cell Count at 15 Minutes Optiflux vs % Change in White Cell Count at 15 Minutes Revaclear; Test type: Superiority; p = 0.534, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 2: Comparison: % Change in White Cell Count at 15 Minutes Optiflux vs % Change in White Cell Count at 15 Minutes ELISIO; Test type: Superiority; p = 0.578, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 3: Comparison: % Change in White Cell Count at 15 Minutes Revaclear vs % Change in White Cell Count at 15 Minutes ELISIO; Test type: Superiority; p = 0.225, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 4: Comparison: % Change in White Cell Count at 30 Minutes Optiflux vs % Change in White Cell Count at 30 Minutes Revaclear; Test type: Superiority; p = 0.125, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 5: Comparison: % Change in White Cell Count at 30 Minutes Optiflux vs % Change in White Cell Count at 30 Minutes ELISIO; Test type: Superiority; p = 0.466, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 6: Comparison: % Change in White Cell Count at 30 Minutes Revaclear vs % Change in White Cell Count at 30 Minutes ELISIO; Test type: Superiority; p = 0.534, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 7: Comparison: % Change in White Cell Count at 60 Minutes Optiflux vs % Change in White Cell Count at 60 Minutes Revaclear; Test type: Superiority; p = 0.584, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 8: Comparison: % Change in White Cell Count at 60 Minutes Optiflux vs % Change in White Cell Count at 60 Minutes ELISIO; Test type: Superiority; p = 0.981, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 9: Comparison: % Change in White Cell Count at 60 Minutes Revaclear vs % Change in White Cell Count at 60 Minutes ELISIO; Test type: Superiority; p = 0.568, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 10: Comparison: % Change in White Cell Count at 240 Minutes Optiflux vs % Change in White Cell Count at 240 Minutes Revaclear; Test type: Superiority; p = 0.240, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 11: Comparison: % Change in White Cell Count at 240 Minutes Optiflux vs % Change in White Cell Count at 240 Minutes ELISIO; Test type: Superiority; p = 0.724, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 20]
Statistical Analysis 12: Comparison: % Change in White Cell Count at 240 Minutes Revaclear vs % Change in White Cell Count at 240 Minutes ELISIO; Test type: Superiority; p = 0.445, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]

7. Primary Outcome: Hemocompatibility as Shown by Platelets for Optiflux, Revaclear, and ELISIO Hemodialysis Dialyzers
Description: Measure of the % change from Baseline for the hemocompatibility marker Platelets for the Optiflux, Revaclear, and ELISIO dialyzers.
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Groups:
- % Change in Platelets at 15 Minutes Optiflux; % Change in Platelets at 15 Minutes Revaclear; % Change in Platelets at 15 Minutes ELISIO: Percent change from baseline at 15 minutes for Platelets.
- % Change in Platelets at 30 Minutes Optiflux; % Change in Platelets at 30 Minutes Revaclear; % Change in Platelets at 30 Minutes ELISIO: Percent change from baseline at 30 minutes for Platelets.
- % Change in Platelets at 60 Minutes Optiflux; % Change in Platelets at 60 Minutes Revaclear; % Change in Platelets at 60 Minutes ELISIO: Percent change from baseline at 60 minutes for Platelets.
- % Change in Platelets at 240 Minutes Optiflux; % Change in Platelets at 240 Minutes Revaclear; % Change in Platelets at 240 Minutes ELISIO: Percent change from baseline at 240 minutes for Platelets.
Arm/Group | % Change in Platelets at 15 Minutes Optiflux | % Change in Platelets at 15 Minutes Revaclear | % Change in Platelets at 15 Minutes ELISIO | % Change in Platelets at 30 Minutes Optiflux | % Change in Platelets at 30 Minutes Revaclear | % Change in Platelets at 30 Minutes ELISIO | % Change in Platelets at 60 Minutes Optiflux | % Change in Platelets at 60 Minutes Revaclear | % Change in Platelets at 60 Minutes ELISIO | % Change in Platelets at 240 Minutes Optiflux | % Change in Platelets at 240 Minutes Revaclear | % Change in Platelets at 240 Minutes ELISIO
Number analyzed (Participants) | 9 | 10 | 9 | 9 | 10 | 9 | 9 | 10 | 9 | 9 | 10 | 9
Percent Change from Baseline | -6.2 (3.9) | -3.1 (4.1) | -3.9 (5.0) | -5.0 (6.2) | -1.5 (4.5) | -9.1 (6.6) | -4.4 (7.8) | -4.8 (5.3) | -7.3 (5.6) | -2.0 (7.5) | 0.7 (12.2) | -1.2 (12.3)
Statistical Analysis 1: Comparison: % Change in Platelets at 15 Minutes Optiflux vs % Change in Platelets at 15 Minutes Revaclear; Test type: Superiority; p = 0.114, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 2: Comparison: % Change in Platelets at 15 Minutes Optiflux vs % Change in Platelets at 15 Minutes ELISIO; Test type: Superiority; p = 0.292, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 3: Comparison: % Change in Platelets at 15 Minutes Revaclear vs % Change in Platelets at 15 Minutes ELISIO; Test type: Superiority; p = 0.714, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 4: Comparison: % Change in Platelets at 30 Minutes Optiflux vs % Change in Platelets at 30 Minutes Revaclear; Test type: Superiority; p = 0.176, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 5: Comparison: % Change in Platelets at 30 Minutes Optiflux vs % Change in Platelets at 30 Minutes ELISIO; Test type: Superiority; p = 0.190, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 6: Comparison: % Change in Platelets at 30 Minutes Revaclear vs % Change in Platelets at 30 Minutes ELISIO; Test type: Superiority; p = -0.009, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 7: Comparison: % Change in Platelets at 60 Minutes Optiflux vs % Change in Platelets at 60 Minutes Revaclear; Test type: Superiority; p = 0.911, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 8: Comparison: % Change in Platelets at 60 Minutes Optiflux vs % Change in Platelets at 60 Minutes ELISIO; Test type: Superiority; p = 0.388, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 9: Comparison: % Change in Platelets at 60 Minutes Revaclear vs % Change in Platelets at 60 Minutes ELISIO; Test type: Superiority; p = 0.337, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 10: Comparison: % Change in Platelets at 240 Minutes Optiflux vs % Change in Platelets at 240 Minutes Revaclear; Test type: Superiority; p = 0.575, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 11: Comparison: % Change in Platelets at 240 Minutes Optiflux vs % Change in Platelets at 240 Minutes ELISIO; Test type: Superiority; p = 0.880, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]
Statistical Analysis 12: Comparison: % Change in Platelets at 240 Minutes Revaclear vs % Change in Platelets at 240 Minutes ELISIO; Test type: Superiority; p = 0.731, t-test, 2 sided; [statistical method as in outcome 1, analysis 20]

ADVERSE EVENTS:
Time Frame: Participant was monitored continuously each of the three dialysis sessions per week over the three week study period.
Description: Adverse events would be comprised of any clinically relevant event during the time the patient was on the study.
Groups:
- Experimental: ELISIO: This group were dialyzed three times in during one week with the ELISO Dialyzer. There were no adverse events during any of the study periods.
- Experimental: Revaclear: This group were dialyzed three times in during one weekwith the Revaclear dialyzer. There were no adverse events during any of the study periods
- Experimental: Optiflux: This group was dialyzed three times in during one weekwith the Optiflux dialyzer. There were no adverse events during any of the study periods
Arm/Group | Experimental: ELISIO | Experimental: Revaclear | Experimental: Optiflux
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-09-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT02433210/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT02433210/SAP_001.pdf